CLINICAL TRIAL: NCT05087680
Title: An Acceptance Based PrEP Intervention to Engage Young Black MSM in the South
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACTPrEP
Record Dates: First submitted 2021-09-13; First posted 2021-10-21 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: HIV Prevention
Keywords: ACT; PrEP

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Control group will include one 30-minute PrEP education session.
  Interventions: Behavioral: Enhanced Standard of Care
- ACTPrEP (Experimental): ACTPrEP will include a 60-minute initial session and 30-minute sessions at 2, 6, and 12 weeks.
  Interventions: Behavioral: ACTPrEP

INTERVENTIONS:
Behavioral: ACTPrEP — ACTPrEP will include a 60-minute initial session and a series of 30-minute follow-up sessions. Sessions will focus on the Thoughts, Emotions, Associations, Memories, and Sensations (TEAMS) relevant to PrEP uptake and adherence.
  Arms: ACTPrEP
Behavioral: Enhanced Standard of Care — Enhanced Standard of Care (ESOC) will include one 30-minute PrEP education session.
  Arms: Control Group

SUMMARY:
Investigators will use a generalized framework for the adaptation of EBIs to inform the development of a brief Acceptance and Commitment Therapy (ACT)-based culturally appropriate pre-exposure prophylaxis (PrEP) intervention tailored to young Black men who have sex with men (YBMSM), named ACTPrEP.

DETAILED DESCRIPTION:
Investigators will use a generalized framework for the adaptation of EBIs to inform the development of a brief Acceptance and Commitment Therapy (ACT)-based culturally appropriate pre-exposure prophylaxis (PrEP) intervention tailored to young Black men who have sex with men (YBMSM), named ACTPrEP.

Specific Aim 1) Gather data from YBMSM (n = 20) and clinic staff (n = 10) through in-depth interviews to assess quantitative measures, intervention design, and experiences most relevant to PrEP engagement.

Specific Aim 2) Develop ACTPrEP utilizing Aim 1 data, working iteratively with experts, and an intervention "run through" with a sample of participants.

CLINICAL TRIAL IS AIM 3 ONLY

Specific Aim 3) Evaluate ACTPrEP. Enroll 66 participants. Primary outcomes will be feasibility (measured by percentage eligible, consented, randomized, and retained) and acceptability (measured by the Client Satisfaction Questionnaire). Secondary outcomes will compare ACTPrEP vs. enhanced standard of care condition (ESOC) on behavior outcomes (uptake, adherence, and PrEP persistence) and possible mediators over the course of 24 weeks. Barriers and facilitators to implementing ACTPrEP will be assessed with post-RCT qualitative interviews using the i-PARIHS framework.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Between 18-34 years old
* Male sex assigned at birth
* Identify as African American/Black
* Not enrolled in another PrEP related study
* Able to give consent
* Not taken PrEP in past 3 months
* Report having sex with a man in the past 3 months
* PrEP-eligible according to CDC guidelines

Exclusion Criteria:

* Participating in another PrEP study
* Unable to provide consent

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
ACTPrEP Feasibility | 12 week visit
  ACTPrEP feasibility is measured by percentage of participants retained in the study.
ACTPrEP Acceptability | 12 week visit
  Acceptability is measured with the Client Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Arnold, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Univeristy of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnold T, Giorlando KK, Barnett AP, Gaudiano BA, Antonaccio CM, Elwy AR, Patrick Edet P, Ward LM, Whiteley L, Bailey S, Rogers BG, Leigland A, Rusley JC, Brown LK. Acceptance-Based Pre-Exposure Prophylaxis Intervention (ACTPrEP) to Engage Young Black Men Who Have Sex With Men in the Southern United States: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 20;14:e65921. doi: 10.2196/65921. PMID 40540736

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT05087680/Prot_SAP_000.pdf